CLINICAL TRIAL: NCT04014517
Title: Effect of Peri-operative Immunonutrition on Recurrence and Infections in Crohn's Disease Patients
Acronym: EPIRIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019-001
Record Dates: First submitted 2019-07-08; First posted 2019-07-10 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Crohn Disease
Keywords: Inflammatory Bowel Diseases; Crohn's Disease; Immunonutrition
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — Standard of Care; Immunonutrition Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator): Standard of Care is represented by the best standard peri-operative treatment already planned for the study population: as for ERAS guidelines, it is represented by fast restoration of liquid and solid diet after surgery (approximately 24 hours after surgery) and pre-operative and post-operative dietary counselling whenever indicated by the surgeon or gastroenterologist
  Interventions: Other: Standard of Care
- Immunonutrition (Experimental): Impact
  Interventions: Dietary Supplement: Immunonutrition

INTERVENTIONS:
Other: Standard of Care — Standard of Care is represented by the best standard peri-operative treatment already planned for the study population: as for ERAS guidelines, it is represented by fast restoration of liquid and solid diet after surgery (approximately 24 hours after surgery) and pre-operative and post-operative dietary counselling whenever indicated by the surgeon or gastroenterologist
  Arms: Standard of Care
Dietary Supplement: Immunonutrition — Impact. Patients will be asked to consume 3 cartons/day of Nestle IMPACT for pre-operative 7 days and 1 carton/day of Nestle IMPACT for post-operative 30 days
  Arms: Immunonutrition

SUMMARY:
This is an interventional randomized ope-label two-arm trial on the peri-operative use of immunonutrition in Crohn's Disease (CD) patients undergoing colorectal elective surgery.The aim of the trial is to assess the effectiveness of immunonutrition therapy in decreasing the rate of post-operative infective complications and 6 months endoscopic disease recurrence.

DETAILED DESCRIPTION:
Crohn's Disease (CD) patients undergoing abdominal surgery are at high risk to develop post-operative surgical and medical infective complications. Infective complications affect almost 24% of patients. Post-surgical disease recurrence afflicts 35-85% of CD patients in the first year after surgery. Immunonutrition has been successfully applied to surgical patients in several randomized trials, demonstrating a decreased rate of post-operative infective complications. The aim of the study is to compare the incidence of surgical and medical post-operative infective complications and six months endoscopic and clinical disease recurrence (DR) in CD patients receiving immunonutrition in the peri-operative setting compared to patients treated as for standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years old, females or males;
* Established Crohn's Disease at the time of surgery indication;
* Patients scheduled for elective open or minimally invasive bowel resection or strictureplasty;
* Patients planned for concomitant perianal surgery for CD-related perianal disease can be included in the study.

Exclusion Criteria:

* Patients < 18 years old;
* Pregnant or breastfeeding women;
* Diagnosis of undetermined colitis;
* Concomitant diagnosis of malignancy;
* Established malnutrition, according to clinical definition, requiring nutritional intervention;
* Patients with more than two criteria for high risk of recurrence among the following: previous abdominal resection, penetrating disease phenotype or active smoking;
* Any condition that, in the opinion of the investigator, can interfere with the consent procedure or the conduction of the trial;
* Patients known to have allergic history to any component of the investigational product;
* Patient with liver and kidney dysfunction (alanine aminotransferase ALT ≥ 2 times the upper limit of normal; total bilirubin TBIL ≥ 2 times the upper limit of normal; creatinine Cr ≥ 2 times the upper limit of normal);
* Patients diagnosed with diabetes or fasting blood glucose≥ 10mmol/L;
* Planned recovery shorter than 48 hours;
* Surgery in emergency setting;
* Any concomitant surgery not related to CD or perianal CD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Post-operative infective complications rate | 30 days post-operatively
  Post-operative infective complications rate (including intra-abdominal septic complications, surgical site infections and medical inflections) will be evaluated with clinical, radiological and molecular analysis
6 months endoscopic recurrence | 6 months post-operatively
  Endoscopic recurrence will be evaluated through colonoscopy with or without biopsies and Rutgeert score. Rutgeert score is an endoscopic risk score intended to predict disease recurrence: it is calculated depending on the number and type of intestinal lesions and consists of five level of disease recurrence risk, from 0 (endoscopic remission) to 4 (advanced disease recurrence).

SECONDARY OUTCOMES:
6 months nutritional status | 6 months post-operatively
  Nutritional status will be evaluated through the Malnutrition Universal Screening Tool (MUST). MUST consists of three different levels, generating a risk predictor ranging from 0 (low risk) to 2 (high risk), considering the calculated Body Mass Index (BMI), the unintentional weight loss and the pathological conditions of the patient.
30 days quality of life | 30 days post-operatively
  Quality of Life will be evaluated trhough the Short-Inflammatory Bowel Disease Quality of Life questionnaire (S-IBDQoL), which is 10-item questionnaire. All items are reported in a 7 point scale, from "all of the time" to "none of the time" (1 = poor health; 7 = good health).
90 days quality of life | 90 days post-operatively
  Quality of Life will be evaluated trhough the Short-Inflammatory Bowel Disease Quality of Life questionnaire (S-IBDQoL), which is 10-item questionnaire. All items are reported in a 7 point scale, from "all of the time" to "none of the time" (1 = poor health; 7 = good health).
6 months quality of life | 6 months post-operatively
  Quality of Life will be evaluated trhough the Short-Inflammatory Bowel Disease Quality of Life questionnaire (S-IBDQoL), which is 10-item questionnaire. All items are reported in a 7 point scale, from "all of the time" to "none of the time" (1 = poor health; 7 = good health).

CONTACTS AND LOCATIONS:
Overall Officials: Antonino Spinelli, MD, PhD, Principal Investigator — Istituto Clinico Humanitas

IPD SHARING:
Plan to Share IPD: No